CLINICAL TRIAL: NCT00258245
Title: A Phase I Study of Arsenic Trioxide and Ascorbic Acid (ATO/AA) in Combination With Low Dose Velcade-Thalidomide-Dexamethasone (VTD) in Relapsed/Refractory Multiple Myeloma (MM)
Brief Title: Arsenic Trioxide and Ascorbic Acid Combined With Bortezomib, Thalidomide, and Dexamethasone in Treating Patients With Relapsed or Refractory Multiple Myeloma or Plasma Cell Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000445464; P30CA022453 (NIH); WSU-D-2869; WSU-HIC-01705M1F
Record Dates: First submitted 2005-11-22; First posted 2005-11-24 (Estimated); Last update posted 2013-04-29 (Estimated); Status verified 2013-04

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage II multiple myeloma; stage III multiple myeloma; refractory multiple myeloma; stage I multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Ascorbic Acid; Arsenic Trioxide; Bortezomib; Dexamethasone; Calcium Dobesilate; dexamethasone 21-phosphate; dexamethasone acetate; Thalidomide; Aspirin; aspirin, aluminum hydroxide, magnesium hydroxide drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bortezomib, AT, Thalidomide, Dexamethasone, Vit C, ASA (Experimental): Bortezomib (Velcade)- 0.7→1.0 mg/m2 IVP d 1, 4, 8, 11; Arsenic Trioxide [AT] (Trisenox)- 0.10→0.15→0.25 mg/kg/dose IVPB days 1, 4, 8, 11; Thalidomide (Thalomid)- 50 mg/day by mouth (PO); Dexamethasone (Decadron)- 40 mg/d IVPB or by mouth (PO) d 1, 4, 8, 11; Ascorbic Acid (Vit C)- 1000 mg IVPB p Arsenic Trioxide (ATO) days 1, 4, 8, 11; Aspirin (ASA)- 325 mg by mouth (PO) every day
  Interventions: Dietary Supplement: ascorbic acid; Drug: arsenic trioxide; Drug: bortezomib; Drug: dexamethasone; Drug: thalidomide; Drug: Aspirin

INTERVENTIONS:
Dietary Supplement: ascorbic acid — Ascorbic Acid (Vit C)- 1000 mg IVPB after Arsenic Trioxide [ATO] days 1, 4, 8, 11
  Other Names: All Day C CR; Ascot; C Complex; C-500; C-500-Gr; C-Time; Cecon; Cemill 1000; Cemill 500; Centrum Singles-Vitamin C; Cevi-Bid; N Ice with Vitamin C; Special C; Sunkist Vitamin C; Vicks Vitamin C Drops; Vitamin C TR
Drug: arsenic trioxide — Arsenic Trioxide (Trisenox)- 0.10→0.15→0.25 mg/kg/dose IVPB days 1, 4, 8, 11
  Other Names: Trisenox®
Drug: bortezomib — Bortezomib (Velcade)- 0.7→1.0 mg/m2 IVP days 1, 4, 8, 11
  Other Names: Velcade®
Drug: dexamethasone — Dexamethasone (Decadron)- 40 mg/days IVPB or PO d 1, 4, 8, 11
  Other Names: Dexasone; Decadron; Diodex; Hexadrol; Maxidex; Dexamethasone Sodium Phosphate; Dexamethasone Acetate
Drug: thalidomide — Thalidomide (Thalomid) - 50 mg/day by mouth (PO)
  Other Names: Thalomid
Drug: Aspirin — Aspirin - 325 mg by mouth (PO) every day
  Other Names: Acuprin 81; Anacin Aspirin Regimen; Ascriptin; Ascriptin Enteric; Aspergum; Aspidrox; Aspir-Low; Aspir-Mox; Aspir-trin; Aspirtab; Bayer Aspirin; Bufferin; Buffex; Easprin; Ecotrin; Ecpirin; Empirin; Entaprin; Entercote; Fasprin; Genacote; Gennin-FC; Genprin; Halfprin; Magnaprin; Med Aspirin; Migralex; Miniprin; Minitabs; Norwich Aspirin; Ridiprin; Sloprin; St. Joseph Aspirin; Uni-Buff; Uni-Tren; Valomag; Zero-Order Release; Zorprin

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as arsenic trioxide and dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Ascorbic acid may help arsenic trioxide work better by making cancer cells more sensitive to the drug. Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Thalidomide may stop the growth of cancer cells by stopping blood flow to the cancer. Giving arsenic trioxide and ascorbic acid together with bortezomib, thalidomide, and dexamethasone may stop the growth of and kill more cancer cells.

PURPOSE: This phase I trial is studying the side effects and best dose of arsenic trioxide when given together with ascorbic acid, bortezomib, thalidomide, and dexamethasone in treating patients with relapsed or refractory multiple myeloma or plasma cell leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the dose-limiting toxicity of arsenic trioxide when given in combination with ascorbic acid, bortezomib, thalidomide, and dexamethasone, particularly in terms of sensory neuropathy, in patients with relapsed or refractory multiple myeloma or plasma cell leukemia.

Secondary

* Determine the overall response rate, complete response rate, and response duration in patients treated with the maximum tolerated dose of this regimen.
* Determine whether the addition of arsenic trioxide and ascorbic acid to the treatment regimen (beginning in course 2) increases NFKB inhibition in these patients during courses 2 and 3 compared to course 1.

OUTLINE: This is a multicenter, dose-escalation study of arsenic trioxide.

* Induction therapy: Patients receive bortezomib IV over 3-5 seconds and dexamethasone IV or orally on days 1, 4, 8, and 11 and oral thalidomide once daily on days 1-21 (course 1). For course 2 and all subsequent courses, patients receive arsenic trioxide IV over 1-2 hours, ascorbic acid IV over 15 minutes, bortezomib IV over 3-5 seconds, and dexamethasone IV or orally on days 1, 4, 8, and 11 and thalidomide once daily on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients who achieve a plateau in response proceed to maintenance therapy.
* Maintenance therapy: Patients receive oral dexamethasone every other day and oral thalidomide once daily in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of arsenic trioxide until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: A total of 24 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed multiple myeloma (MM) or plasma cell leukemia meeting 1 of the following criteria:

  * Relapsed or refractory disease after treatment with prior effective therapy
  * Exhibited < a partial response to the last therapy
* Measurable disease, defined by 1 of the following:

  * Serum M protein ≥ 1.0 g/dL
  * Urine M-protein ≥ 500 mg/24 hours
  * Plasmacytoma with bidimensional measurements on CT scan or MRI (each axis ≥ 1 cm)
* Previously treated with ≥ 1 induction chemotherapy regimen for MM
* No known CNS involvement by multiple myeloma

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod or SWOG 0-2 OR
* Karnofsky 60-100%

Life expectancy

* More than 12 weeks

Hematopoietic

* WBC ≥ 1,500/mm^3
* Absolute neutrophil count ≥ 1,000/mm^3
* Platelet count ≥ 80,000/mm^3
* Hemoglobin ≥ 8.5 g/dL
* No history of heparin-induced thrombocytopenia

  * Low blood counts allowed if marrow is heavily infiltrated by multiple myeloma

Hepatic

* Bilirubin ≤ 1.5 times upper limit normal (ULN)
* AST and ALT ≤ 2.5 times ULN

Renal

* Creatinine ≤ 2.5 mg/dL

Cardiovascular

* QTc < 480 msec on EKG in the presence of serum potassium ≥ 4.0 mEq/dL and serum magnesium ≥ 1.8 mg/dL
* LVEF ≥ 55% by ECHO or MUGA
* No prior deep vein thrombosis, unless on concurrent anticoagulation
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No history of ventricular arrhythmia

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after completion of study treatment
* No history of allergic reactions or severe adverse reactions attributed to compounds of similar chemical or biological composition to study drugs
* No other malignancy in the past 2 years except adequately treated nonmelanoma skin cancer or carcinoma in situ of the cervix
* No peripheral neuropathy ≥ grade 2
* No ongoing or active infection requiring IV antibiotics
* No psychiatric illness or social situation that would preclude study compliance
* No other uncontrolled illness
* Controlled HIV disease allowed as long as there are no associated comorbid complications
* No active peptic ulcer disease
* No other condition that would confer a high risk of bleeding complications

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 4 weeks since prior thalidomide or lenalidomide for MM
* Prior autologous or allogeneic stem cell transplant for MM allowed
* Concurrent hematopoietic growth factors (e.g., epoetin alfa, filgrastim [G-CSF]) for MM allowed

Chemotherapy

* See Disease Characteristics
* More than 4 weeks since prior arsenic trioxide for MM

Endocrine therapy

* More than 4 weeks since prior corticosteroids for MM

Radiotherapy

* More than 4 weeks since prior therapeutic radiotherapy (e.g., to plasmacytomas)

  * Palliative radiotherapy for painful symptomatic lytic skeletal lesions allowed within the past 4 weeks

Surgery

* Not specified

Other

* More than 4 weeks since prior cytotoxic agents or other therapy (e.g., bortezomib) for MM
* More than 30 days (or 5 half-lives) since prior investigational agents
* Concurrent bisphosphonates for MM allowed
* No other concurrent anticancer therapy
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2005-05; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
To determine if arsenic trioxide and ascorbic acid at doses up to 0.25 mg/mg/dose can be given in combination with reduced-dose dexamethasone, bortezomib and thalidomide without dose limiting toxicity, especially sensory neuropathies. | Days 1, 4, 8 & 11 of each 21 day cycle

SECONDARY OUTCOMES:
Estimate the Overall Response Rate (ORR), Complete Response Rate (CRR), and Response Duration (RD) in patients treated with the Maximally Tolerated Dose (MTD) of this regimen. | at cycle 2 and 6 weeks after
Determine if addition of Arsenic Trioxide[AT]/Ascorbic Acid (Vit C)[AA] starting in cycle 2 of treatment increases NF-kappa-B [NFKB] inhibition in cycles 2 and 3 compared to cycle 1. | At baseline and 1 hour after the first dose of Bortezomib in cycles 1, 2, and 3
  Peripheral blood samples are to be obtained at baseline, and 1 hour after the first dose of Bortezomib in cycles 1, 2, and 3 for Pharmacodynamic studies

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A. Zonder, MD, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States